CLINICAL TRIAL: NCT03941223
Title: A Prospective, Randomized Comparison Between Paravertebral and Pectoral Nerve Block on Postoperative Pain, Persistent Post Surgical Pain and Cancer Recurrence After Mastectomy
Brief Title: Regional Anesthesia for Breast Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study never started
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Breastblock
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: breast cancer, regional anesthesia, cancer recurrence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pectoral PECS II block (Experimental): Ultrasound-guided PECS II block with ropivacaine 0.75% 20 ml (patients N = 75) + Parasternal ultrasound-guided block at T2, T4 levels with ropivacaine 0.375% 10 ml
  Interventions: Procedure: PECSII and paravertebral blocks
- Paravertebral nerve block (Active Comparator): Ultrasound-guided paravertebral block with ropivacaine 0.75% 20 ml at T1-T2 and T3-T4 levels (10 ml each) (patients N = 75)
  Interventions: Procedure: PECSII and paravertebral blocks

INTERVENTIONS:
Procedure: PECSII and paravertebral blocks — Regional anesthesia for mastectomy outcomes

SUMMARY:
Patients scheduled for mastecotmy will be randomized to receive either an ultrasound-guided double space paravertebral block or a PECSII + parasternal block. In both groups, blocks will be performed with 20 ml of ropivacaine 0.75%, plus ropivacaine 0.375% 10 ml for parasternal block only.

Postoperative, all patients will receive a morphine PCA. They will follow at 6, 12, 24 months for persistent postoperative surgical pain (PPSP) and cancer recurrence.

DETAILED DESCRIPTION:
Patients scheduled for mastecotmy with or without axillary dissection, will be randomized to receive preoperative either an ultrasound-guided double space paravertebral block or a PECSII + parasternal block. In both groups, blocks will be performed with 20 ml of ropivacaine 0.75%, plus ropivacaine 0.375% 10 ml for parasternal block only.

All the patients also received a general anesthesia induced by propofol and esmeron for endotracheal intubation and desflurane for maintaining.

Sensory block by ice and pinprick test application and maximum spread after 40' from LA injection will be registered.

Postoperative, all patients will receive a morphine PCA, ketorolac 30 mg/12h and paracetamol 1g each 8h.

Morphine consumption will be registered. Patients will follow at 6, 12, 24 months for persistent postoperative surgical pain (PPSP) and cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for radical mastectomy for cancer.
* age > 18 y-o
* Written informed consent

Exclusion Criteria:

* Bilateral surgery
* Opioids user
* BMI > 35
* Postoperative Intensive care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Morphine requirement | 1 day
  Morphine self-administered by a patient controlled device

SECONDARY OUTCOMES:
postoperative pain | 2 days
  Pain reporter by a numerical rating scale (NRS) 0-10 (0=no pain, 10=the worst imaginable pain) postoperatively
Persistent Postsurgical pain (PPSP) | 2 years
  Pain reported by a a numerical rating scale (NRS) 0-10 (0=no pain, 10=the worst imaginable pain) in the follow up
cancer recurrence | 2 years
  Incidence of cancer recurrence

CONTACTS AND LOCATIONS:
Overall Officials: gianluca cappelleri, MD, Principal Investigator — AUSL IRCCS Reggio Emilia, Italy
Locations (1):
- AUSL IRCCS Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No